CLINICAL TRIAL: NCT06585176
Title: Epidemiological Studies and Risk Factor Analysis of Gastroesophageal Reflux Diseases in Xiamen City: a Cross-sectional Study
Brief Title: Epidemiological Studies and Risk Factor Analysis of GERD in Xiamen City
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Hospital (Xiamen), Fudan University (Other)
Responsible Party: Principal Investigator, Zhuyucheng, Deputy Chief Physician, Zhongshan Hospital (Xiamen), Fudan University
Other Study IDs: ZYC-GERD2024
Record Dates: First submitted 2024-08-26; First posted 2024-09-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Reflux Disease; Epidemiology; Risk Factors
Keywords: Gastroesophageal reflux diseases; Barrett esophageal
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastroesophageal Reflux Disease: Gastroesophageal reflux disease (GERD) is a gastrointestinal motility disorder that results from the reflux of stomach contents into the esophagus or oral cavity resulting in symptoms or complications.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This concerns a natural history study. No interventions will be used.

SUMMARY:
Gastroesophageal Reflux Disease (GERD) is a condition characterized by the reflux of gastric and duodenal contents into the esophagus, primarily manifested by symptoms such as acid regurgitation and heartburn. GERD significantly affects patients' daily lives and health-related quality of life. Prolonged gastroesophageal reflux can lead to repeated irritation of the esophageal mucosa by gastric acid and acidic gastric contents, resulting in the replacement of normal squamous epithelium in the lower esophagus with metaplastic columnar epithelium. This pathological change, known as Barrett's Esophagus (BE), is considered a precancerous lesion for esophageal adenocarcinoma.

DETAILED DESCRIPTION:
GERD is a common gastrointestinal disorder with numerous risk factors that negatively impact patients' quality of life. Abnormal psychological conditions may influence various aspects of GERD, including its onset, diagnosis, treatment, and prognosis. The incidence and risk factors of GERD vary in different countries or regions. Currently, there is a lack of unified national epidemiological data on GERD in China. Conducting epidemiological studies on GERD in China to identify risk factors and develop prevention and treatment measures tailored to the country's or specific regions' circumstances is crucial for reducing the incidence of GERD and improving patients' quality of life.

In the context of the modern biomedical model of "biopsychosocial" health, actively researching the psychological conditions of patients, while also addressing their physical ailments and providing psychological treatment, emphasizes holistic care. This approach may comprehensively alleviate disease symptoms and enhance quality of life, potentially leading to new breakthroughs in the treatment of GERD.

Based on this, a specialized cohort for gastroesophageal reflux disease will be established, along with multicenter epidemiological and clinical research in the Xiamen area. This initiative will help clarify the etiology of GERD and provide firsthand resources for evidence-based prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients had experienced typical reflux symptoms, i.e., mild heartburn and/or regurgitation symptoms, for at least 2 days per week or moderate/severe reflux symptoms for more than 1 day per week during the previous 3 months and had upper endoscopy examinations in the previous month.
* Cooperate with the questionnaire survey.
* Volunteer and sign the informed consent form.
* Permanent residents in Xiamen.

Exclusion Criteria:

* Malignant tumor.
* Partial or total gastrectomy.
* Failing to cooperate with the investigation because of the factors such as education level and language intelligence disorder, etc.
* Patients with severe heart, lung, kidney, liver, blood, nerve, endocrine and mental system diseases.
* Patients with mental retardation, etc.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastroesophageal reflux disease (GERD) is a common digestive disorder in the general population that primarily affects the esophagus and gastro-duodenum. Due to its prevalence, GERD has a significant impact on quality of life and healthcare costs.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of GERD in Xiamen city | 3 months.
  Gastroesophageal reflux disease (GERD) is the most prevalent gastrointestinal disorder in the world. In this study, we will study the incidence of GERD in Xiamen city.
The percentage of reflux esophagitis | 3 months.
  The percentage of participants diagnosed with reflux esophagitis using endoscopy among patients with baseline symptoms.
The percentage of Barrett esophagus | 3 months.
  The percentage of paticipants diagnosed with pathological Barrett esophagus using endoscopy monitoring among patients with baseline symptom in gastroenterology department will be calculated.

SECONDARY OUTCOMES:
The life quality of GERD patients who were diagnosed by endoscopy | 3 months.
  The life quality of GERD patients with different main symptoms before PPI test will be measured via the 50-item short form health survey , in which higher scores mean a better quality of life.
The sensitivity of GERD-Q for diagnosis of GERD | 3 months.
  The sensitivity of GERD-Q for the diagnosis of GERD in patients with typical or atypical reflux symptoms will be calculated. The presence of reflux esophagitis on upper endoscopy and/or pathological acid reflux on 24-hour pH monitoring are considered as the gold standard for the diagnosis of GERD.
The specificity of GERD-Q for diagnosis of GERD | 3 months.
  The specificity of GERD-Q for the diagnosis of GERD in patients with typical or atypical reflux symptoms will be calculated. The presence of reflux esophagitis on upper endoscopy and/or pathological acid reflux on 24-hour pH monitoring are considered as the gold standard for the diagnosis of GERD.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Doctor, Study Chair — Zhongshan Hospital (Xiamen), Fudan University
Locations (1):
- Zhongshan Hospital (Xiamen), Fudan University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Katz PO, Dunbar KB, Schnoll-Sussman FH, Greer KB, Yadlapati R, Spechler SJ. ACG Clinical Guideline for the Diagnosis and Management of Gastroesophageal Reflux Disease. Am J Gastroenterol. 2022 Jan 1;117(1):27-56. doi: 10.14309/ajg.0000000000001538. PMID 34807007
- [Result] Chen Y, Sun X, Fan W, Yu J, Wang P, Liu D, Song M, Liu S, Zuo X, Zhang R, Hou Y, Han S, Li Y, Zhang J, Li X, Ke M, Fang X. Differences in Dietary and Lifestyle Triggers between Non-Erosive Reflux Disease and Reflux Esophagitis-A Multicenter Cross-Sectional Survey in China. Nutrients. 2023 Jul 31;15(15):3400. doi: 10.3390/nu15153400. PMID 37571337